CLINICAL TRIAL: NCT02207920
Title: A Phase 1b Clinical Trial to Evaluate the Safety and Immunogenicity of Different Combinations of DNA-HIV-PT123 and AIDSVAX® B/E in Healthy, HIV Uninfected Adult Participants
Brief Title: Evaluating the Safety and Immune Response to Different Combinations of the DNA-HIV-PT123 and AIDSVAX® B/E Vaccines in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 105; 11986 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX B-E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): At study entry and Month 1, participants will receive placebo for DNA-HIV-PT123 in their left deltoid and AIDSVAX B/E in their right deltoid.
  At Months 3 and 6, participants will receive DNA-HIV-PT123 in their left deltoid and placebo for AIDSVAX B/E in their right deltoid.
  Interventions: Biological: AIDSVAX B/E Vaccine; Biological: DNA-HIV-PT123 Vaccine; Biological: Placebo for DNA-HIV-PT123; Biological: Placebo for AIDSVAX B/E
- Group 2 (Experimental): At study entry and Month 1, participants will receive DNA-HIV-PT123 in their left deltoid and placebo for AIDSVAX B/E in their right deltoid.
  At Months 3 and 6, participants will receive placebo for DNA-HIV-PT123 in their left deltoid and AIDSVAX B/E in their right deltoid.
  Interventions: Biological: AIDSVAX B/E Vaccine; Biological: DNA-HIV-PT123 Vaccine; Biological: Placebo for DNA-HIV-PT123; Biological: Placebo for AIDSVAX B/E
- Group 3 (Experimental): At study entry and Month 1, participants will receive DNA-HIV-PT123 in their left deltoid and placebo for AIDSVAX B/E in their right deltoid.
  At Months 3 and 6, participants will receive DNA-HIV-PT123 in their left deltoid and AIDSVAX B/E in their right deltoid.
  Interventions: Biological: AIDSVAX B/E Vaccine; Biological: DNA-HIV-PT123 Vaccine; Biological: Placebo for AIDSVAX B/E
- Group 4 (Experimental): At study entry and Months 1, 3, and 6, participants will receive DNA-HIV-PT123 in their left deltoid and AIDSVAX B/E in their right deltoid.
  Interventions: Biological: AIDSVAX B/E Vaccine; Biological: DNA-HIV-PT123 Vaccine

INTERVENTIONS:
Biological: AIDSVAX B/E Vaccine — 600 mcg/mL to be administered as 1 mL intramuscular (IM) injection
Biological: DNA-HIV-PT123 Vaccine — 4 mg/mL to be administered as 1 mL IM injection
Biological: Placebo for DNA-HIV-PT123 — Sodium chloride for injection USP, 0.9%; administered as 1 mL IM injection
  Arms: Group 1; Group 2
Biological: Placebo for AIDSVAX B/E — Sodium chloride for injection USP, 0.9%; administered as 1 mL IM injection
  Arms: Group 1; Group 2; Group 3

SUMMARY:
This study will evaluate the safety, tolerability, and immune response to different combinations of two experimental HIV vaccines-the DNA-HIV-PT123 vaccine and the AIDSVAX® B/E vaccine-in healthy adults who are not infected with HIV.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of the combination of two different experimental HIV vaccines-the DNA-HIV-PT123 vaccine and the AIDSVAX® B/E vaccine-administered in different sequences or simultaneously, in healthy adults who are not infected with HIV.

Participants will be randomly assigned to four groups. Depending on which group participants are in, they will receive different combinations of the DNA-HIV-PT123 vaccine, the AIDSVAX® B/E vaccine, a placebo for DNA-HIV-PT123 vaccine, and/or a placebo for AIDSVAX® B/E vaccine. Study visits will occur at study entry, Week 2, and Months 1, 1.5, 3, 3.5, 6, 6.5, 9, and 12. All participants will receive their assigned combinations of vaccines at study entry and Months 1, 3, and 6. At each vaccination visit, participants will receive one injection in each upper arm. Following each vaccination, participants will remain in the clinic for 30 minutes for monitoring. All study visits will include a physical examination, HIV risk reduction counseling, and questionnaires and assessments. Select study visits will also include a urine collection, a blood collection, a pregnancy test for participants who were born female, and HIV testing and counseling.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study; completes a questionnaire prior to first vaccination, with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent before the last required protocol clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit

Laboratory Inclusion Values

Hemogram/Complete Blood Count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female; greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT) less than 1.25 times the institutional upper limit of normal (IULN) and creatinine less than or equal to IULN

Virology

* Negative HIV-1 and -2 blood test: participants must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA)
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus (anti-HCV) Abs, or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cell levels within institutional normal range)

Reproductive Status

* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy with bilateral oophorectomy (verified by medical records) are not required to undergo pregnancy testing.
* Reproductive status: a participant who was born female must:

  * Agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit;
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent. More information on this criterion is available in the protocol.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with 2 or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, or known hyperlipidemia
* Intent to participate in another study of an investigational research agent before the last required protocol clinic visit
* Pregnant or breastfeeding

Vaccines and Other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For participants who have received control/placebo in an HIV vaccine trial, the HVTN 105 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by FDA. For participants who have received control/placebo in an experimental vaccine trial, the HVTN 105 PSRT will determine eligibility on a case-by-case basis. For participants who have received an experimental vaccine(s) more than 5 years ago, eligibility for enrollment will be determined by the HVTN 105 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses less than 2 mg/kg/day and length of therapy less than 11 days, with completion at least 30 days prior to enrollment)
* Serious adverse reactions to vaccines, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child)
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease (Not excluded: mild, well-controlled psoriasis)
* Immunodeficiency

Clinically Significant Medical Conditions

* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion is available in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma other than mild or moderate, well-controlled asthma. More information on this criterion is available in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* Hypertension:

  * If a participant has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these participants, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a participant has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded: participant who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: history of seizure(s) within the past 3 years. Also exclude if participant has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of local and systemic reactogenicity signs and symptoms | Measured through Month 12
Laboratory measure of safety: measurement of complete blood count (CBC) | Measured through Month 12
  Including differential and platelets
Laboratory measure of safety: measurement of alanine aminotransferase (ALT) | Measured through Month 12
Laboratory measure of safety: measurement of creatinine | Measured through Month 12
Frequency of adverse events (AEs) | Measured through Month 12
Frequency of serious adverse events (SAEs) | Measured through Month 12
HIV-specific binding antibody (Ab) response as assessed by binding Ab multiplex assay | Measured 2 weeks after the 4th vaccination
Response rate and magnitude of CD4 T cell responses as assessed by intracellular cytokine staining (ICS) assays | Measured 2 weeks after the 4th vaccination
Response rate and magnitude of CD8 T cell responses as assessed by ICS assays | Measured 2 weeks after the 4th vaccination

SECONDARY OUTCOMES:
Neutralizing antibody (nAb) magnitude and breadth against tier 1 and tier 2 HIV-1 isolates as assessed by area under the magnitude-breadth curves | Measured 2 weeks after the 4th vaccination
Measurement of HIV-specific Ab and T-cell responses | Measured 6 months after the 4th vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Michael Keefer, Study Chair — University of Rochester
Locations (7):
- United States (7):
  - Bridge HIV CRS, San Francisco, California
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Basu M, Fucile C, Piepenbrink MS, Bunce CA, Man LX, Liesveld J, Rosenberg AF, Keefer MC, Kobie JJ. Mixed Origins: HIV gp120-Specific Memory Develops from Pre-Existing Memory and Naive B Cells Following Vaccination in Humans. AIDS Res Hum Retroviruses. 2023 Jul;39(7):350-366. doi: 10.1089/AID.2022.0104. Epub 2023 Mar 22. PMID 36762930
- [Derived] Fischinger S, Cizmeci D, Deng D, Grant SP, Frahm N, McElrath J, Fuchs J, Bart PA, Pantaleo G, Keefer M, O Hahn W, Rouphael N, Churchyard G, Moodie Z, Donastorg Y, Streeck H, Alter G. Sequence and vector shapes vaccine induced antibody effector functions in HIV vaccine trials. PLoS Pathog. 2021 Nov 29;17(11):e1010016. doi: 10.1371/journal.ppat.1010016. eCollection 2021 Nov. PMID 34843602
- [Derived] Basu M, Piepenbrink MS, Francois C, Roche F, Zheng B, Spencer DA, Hessell AJ, Fucile CF, Rosenberg AF, Bunce CA, Liesveld J, Keefer MC, Kobie JJ. Persistence of HIV-1 Env-Specific Plasmablast Lineages in Plasma Cells after Vaccination in Humans. Cell Rep Med. 2020 May 19;1(2):100015. doi: 10.1016/j.xcrm.2020.100015. PMID 32577626
- [Derived] Rouphael NG, Morgan C, Li SS, Jensen R, Sanchez B, Karuna S, Swann E, Sobieszczyk ME, Frank I, Wilson GJ, Tieu HV, Maenza J, Norwood A, Kobie J, Sinangil F, Pantaleo G, Ding S, McElrath MJ, De Rosa SC, Montefiori DC, Ferrari G, Tomaras GD, Keefer MC; HVTN 105 Protocol Team and the NIAID HIV Vaccine Trials Network. DNA priming and gp120 boosting induces HIV-specific antibodies in a randomized clinical trial. J Clin Invest. 2019 Nov 1;129(11):4769-4785. doi: 10.1172/JCI128699. PMID 31566579